CLINICAL TRIAL: NCT04083989
Title: Adolescent Inpatients With Anorexia Nervosa: Changes in Heart Rate Variability, Body Warmth and Eating Disorder Features - a Prospective Controlled Study
Brief Title: Investigation of Psycho-Physiological Parameters in Adolescent Inpatients With Anorexia Nervosa
Status: Completed | Type: Observational
Sponsor: ARCIM Institute Academic Research in Complementary and Integrative Medicine (Other)
Collaborators: Die Filderklinik, Filderstadt, Germany (Unknown)
Responsible Party: Sponsor
Other Study IDs: ANS_01
Record Dates: First submitted 2019-09-05; First posted 2019-09-10 (Actual); Last update posted 2019-09-10 (Actual); Status verified 2019-09

CONDITIONS: Anorexia Nervosa
Keywords: Anorexia nervosa; Eating disorder; Adolescents; Inpatient treatment; Integrative medicine; Anthroposophic medicine; Heart rate variability; Thermography
MeSH Terms: conditions — Anorexia Nervosa; Feeding and Eating Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Multimodal treatment for AN: Adolescent patients with AN attending an integrative medicine-based inpatient treatment program
  Interventions: Other: Integrative medicine-based multimodal treatment
- Healthy controls: Healthy volunteers assessed once to collect comparative data

INTERVENTIONS:
Other: Integrative medicine-based multimodal treatment — Multimodal inpatient treatment program based on anthroposophic medicine, including individual and group psychotherapy, family therapy, art therapies and specific nursing applications such as embrocations, rhythmical massage and oil dispersion baths.
  Groups: Multimodal treatment for AN

SUMMARY:
A study to assess changes in mental and physical symptoms in adolescent inpatients with anorexia nervosa, a severe eating disorder.

DETAILED DESCRIPTION:
This is a prospective controlled trial to assess changes in psycho-physiological parameters, including eating disorder features (drive for thinness, body dissatisfaction) and comorbid symptoms such as anxiety, depression and quality of life as well as heart rate variability, body warmth and BMI in adolescent inpatients with anorexia nervosa. Parameters were assessed at admission, six weeks after admission and three months thereafter and compared to reference values of healthy controls.

ELIGIBILITY:
Inclusion Criteria:

* Age 11-18 years
* Restrictive subtype of adolescent AN
* Fulfilling the AN diagnostic criteria of the Diagnostic and Statistical Manual of Mental Disorders (DSM-IV and V)
* Admitted to the Filderklinik for inpatient treatment

Exclusion Criteria:

* Patients diagnosed with the binge-purge subtype of adolescent AN or with other eating disorders
* Healthy controls: BMI beyond the defined norm for their age group
* Healthy controls: acute or chronic disorders including psychiatric disorders, heart defects, cardiac arrhythmia, other disorders requiring medication

Ages: 11 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Adolescent patients with Anorexia Nervosa who are admitted to the Filderklinik's ward for eating disorders to attend a specific inpatient treatment program based on anthroposophic medicine
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2013-05-01 (Actual); Primary Completion 2014-10-09 (Actual); Study Completion 2014-10-09 (Actual)

PRIMARY OUTCOMES:
Change in Drive for Thinness | At admission (timepoint 1, t1), six weeks after admission (t2), and three months after t2 (t3)
  Assessed with the 7-item subscale Drive for Thinness of the self-reporting Eating Disorder Inventory-2 at admission to the hospital (t1), six weeks after admission (t2) and three months after t2 (t3)
Change in Body Dissatisfaction | At admission (t1), six weeks after admission (t2), and three months after t2 (t3)
  Assessed with the 9-item subscale Body Dissatisfaction of the self-reporting Eating Disorder Inventory-2 at admission to the hospital (t1), six weeks after admission (t2) and three months after t2 (t3)

SECONDARY OUTCOMES:
Anxiety | At admission (t1), six weeks after admission (t2), and three months after t2 (t3)
  Assessed with the 7-item subscale Anxiety of the self-reporting Hospital Anxiety and Depression Scale at admission to the hospital (t1), six weeks after admission (t2) and three months after t2 (t3)
Depression | At admission (t1), six weeks after admission (t2), and three months after t2 (t3)
  Assessed with the 7-item subscale Depression of the self-reporting Hospital Anxiety and Depression Scale at admission to the hospital (t1), six weeks after admission (t2) and three months after t2 (t3)
SF-12 physical | At admission (t1), six weeks after admission (t2), and three months after t2 (t3)
  Physical health-related quality of life, assessed with the 6-item subscale Physical Health of the self-reporting Health-Related Quality of Life Questionnaire (SF-12) at admission to the hospital (t1), six weeks after admission (t2) and three months after t2 (t3)
SF-12 mental | At admission (t1), six weeks after admission (t2), and three months after t2 (t3)
  Mental health-related quality of life, assessed with the 6-item subscale Mental Health of the self-reporting Health-Related Quality of Life Questionnaire (SF-12) at admission to the hospital (t1), six weeks after admission (t2) and three months after t2 (t3)
SF-12 global | At admission (t1), six weeks after admission (t2), and three months after t2 (t3)
  Overall health-related quality of life, assessed with the self-reporting 12-item Health-Related Quality of Life Questionnaire (SF-12 sum-score) at admission to the hospital (t1), six weeks after admission (t2) and three months after t2 (t3)
Weight gain | At admission (t1), six weeks after admission (t2), and three months after t2 (t3)
  Change in BMI (kg/m2) based on body weight measurements taken at admission to the hospital (t1), six weeks after admission (t2) and three months after t2 (t3)
Heart rate | At admission (t1), six weeks after admission (t2), and three months after t2 (t3)
  Heart rate (beats/min), derived from 24h ECG recordings
Heart rate variability: SDNN | At admission (t1), six weeks after admission (t2), and three months after t2 (t3)
  Standard deviation of normal to normal (NN) intervals (ms), derived from 24h ECG recordings
Body warmth | At admission (t1), six weeks after admission (t2), and three months after t2 (t3)
  Body surface temperature (°C) at the inner canthi of both eyes, measured with high-resolution infrared thermography at admission (t1), six weeks after admission (t2) and three months after t2 (t3)

CONTACTS AND LOCATIONS:
Locations (1):
- Die Filderklinik, Filderstadt, Baden-Wurttemberg, Germany